CLINICAL TRIAL: NCT01839942
Title: Recurrence and Patient Satisfaction After Laparoscopic Hernia Repair With Intraperitoneal Onlay-mesh (IPOM)
Acronym: SGChirIPOM
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Sascha Müller, Attending physician, Cantonal Hospital of St. Gallen
Other Study IDs: SGChirIPOM
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Ventral Hernia; Recurrent Ventral Hernia
Keywords: Hernia, Ventral
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- no gap closure: no hernia gap closure
- extracorporal gap closure: extracorporal hernia gap closure
  extracorporal suturing of gap
  Interventions: Procedure: hernia gap closure; Procedure: extracorporal suturing of gap
- intracorporal gap closure: intracorporal hernia gap closure
  Interventions: Procedure: hernia gap closure

INTERVENTIONS:
Procedure: hernia gap closure — type of gap closure during laparoscopic repair of a ventral hernia: none, extracorporal, intracorporal
  Groups: extracorporal gap closure; intracorporal gap closure
Procedure: extracorporal suturing of gap — ventral hernia gap is sutured extracorporally
  Groups: extracorporal gap closure

SUMMARY:
For laparoscopic ventral hernia repair, the technique to close the hernia gap is not well established. Mainly three techniques are currently applied:

* no closure at all
* extracorporal suturing of the gap
* intracorporal suturing of the gap

All three techniques have been applied at our hospital. Patients who received laparoscopic hernia repair between 2006 and 2011 will be identified from the patient database and will be contacted by phone to inquire about the outcome and the satisfaction of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* hernia repair between 2006 and 2011
* laparoscopic hernia repair using intraperitoneal onlay-mesh (IPOM)
* patient agrees to be surveyed by phone

Exclusion Criteria:

* Patient rejects participation in survey
* patient already rejected use of his/her data for research purposes at admittance to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after laparoscopic repair of a ventral hernia (including recurrent hernias)
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | 7 years
  Hernia recurrence at the time of phone survey (2 - 7 years after surgery)

SECONDARY OUTCOMES:
Time to recurrence | 7 years
  time from surgery to hernia recurrence
Patient satisfaction | 2 - 7 years after surgery
  questionnaire with 4 items and 5 step Likert scales

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Müller, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital St.Gallen, Sankt Gallen, Switzerland